CLINICAL TRIAL: NCT03984214
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial to Investigate the Efficacy and Safety of Dronabinol in the Improvement of ChemOthErapy-induced and Tumor-Related Symptoms in Patients With Locally Advanced or Metastatic Pancreatic Cancer During First-line Chemotherapy (DIsCOvER)
Brief Title: Efficacy and Safety of Dronabinol in the Improvement of Chemotherapy-induced and Tumor-related Symptoms in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Medical University of Graz (Other); Unidata Geodesign (Unknown); Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGMT_DISCOVER
Record Dates: First submitted 2019-05-28; First posted 2019-06-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer Non-resectable; Chemotherapy-induced Nausea and Vomiting; Pancreatic Cancer Metastatic
Keywords: Dronabinol; THC; Placebo; Pancreatic Cancer; Chemotherapy-induced Nausea and Vomiting; Tumor related symptoms; Quality of life; EORTC QLQ-C30; FOLFIRINOX; Abraxane; Gemcitabine
MeSH Terms: conditions — Vomiting; Pancreatic Neoplasms | interventions — Dronabinol; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol (Active Comparator): BX-1 contains 25 mg dronabinol/ml (2.5% delta-9-trans-tetrahydrocannabinol = THC), oral solution; three applications per day from 2.5 mg (3 x 1 droplet) up to 30 mg (3 x 12 droplets)
  Interventions: Drug: Dronabinol in Oral Dosage Form
- Placebo (Placebo Comparator): Placebo: oral solution with cannabis flavor without active substance and otherwise identical to active comparator, three applications per day from 3 x 1 droplet up to 3 x 12 droplets
  Interventions: Drug: Placebo in Oral Dosage Form

INTERVENTIONS:
Drug: Dronabinol in Oral Dosage Form — Titration period for 4 weeks: titration according to tolerability from 2.5 mg (3 x 1 droplet) up to 30 mg (3 x 12 droplets) per day; dose increased by 2.5 mg (3 x 1 droplet) every other day Maintenance period for 12 weeks: individually tolerated maximum dose (up to 30 mg ≙ 3 x 12 droplets) at end of titration period will be continued for maintenance treatment Tapering period for 2 weeks: dose is decreased every other day by 5 mg (3 x 2 droplets) Safety follow-up: 4 weeks after end of treatment
  Other Names: BX-1
  Arms: Dronabinol
Drug: Placebo in Oral Dosage Form — Titration period for 4 weeks: titration according to tolerability from 3 x 1 droplet up to 3 x 12 droplets per day; dose increased by 3 x 1 droplet every other day Maintenance period for 12 weeks: individually tolerated maximum dose (up to 3 x 12 droplets) at end of titration period will be continued for maintenance treatment Tapering period for 2 weeks: dose is decreased every other day by 3 x 2 droplets Safety follow-up: 4 weeks after end of treatment
  Arms: Placebo

SUMMARY:
Aim of this phase III trial is to investigate the efficacy and safety of dronabinol (orally administered tetrahydrocannabinol (THC)) as adjuvant therapy to first-line standard chemotherapy in patients with metastatic pancreatic cancer for improvement of chemotherapy- and tumor-related symptoms applicated by individual titration up to the maximum tolerated dose.

DETAILED DESCRIPTION:
Patients with pancreatic cancer suffer from multiple symptoms related to the tumor itself or induced by the chemotherapy. The available supportive therapy is still not able to relief all symptoms that are caused by the malignancy itself as well as by the antineoplastic therapy.

Additionally, anorexia and weight loss, that often result in increased morbidity and mortality in this patient population as well as in psycho-social burden and suffering in patients and their relatives, are unmet needs in pancreatic cancer patients.

Therapeutic approaches focus on treating the malignancy itself, additional nutritional support and physical examination might prevent patients from further side effects such as sarcopenia.

During the last decades a number of appetite-modulating drugs have been under clinical investigation. A number of studies focused on the endocannabinoid system, which is involved amongst others in appetite-modulating, antiemetic, analgesic and anti-inflammatory processes.

As dronabinol is already used as magistral formulation, its beneficial effect has often been observed in these patients in the clinical routine, especially in patients with therapy-refractory nausea and emesis. Due to its broad efficacy it might be of benefit for patients suffering from malignancy. Thus, investigators want to evaluate the efficacy of dronabinol in the improvement of chemotherapy-induced and tumor-related symptoms in advanced pancreatic patients during systemic first-line chemotherapy. However, data on optimal dosage are conflicting yet.

In detail, investigators want to study whether dronabinol has a positive influence on quality of life and whether symptoms caused by the tumor or by the chemotherapy itself might be palliated by dronabinol. Beneficial and potential harmful side effects and the personal perception of advanced pancreatic cancer patients will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥18
* Patients with diagnosis of locally advanced, inoperable or metastatic pancreatic cancer, eligible for first-line chemotherapy with FOLFIRINOX or gemcitabine+Abraxane®
* According to investigator life expectancy of > 4 months at screening
* Female patients must either be post-menopausal or surgically sterilized or use a highly effective method of birth control (hormonal contraceptives, intra-uterine devices, or diaphragms with spermicide) for the duration of the study and/or must have a negative pregnancy test (female patients with childbearing potential only)
* Willing and able to provide written informed consent.
* Written informed consent given prior to any trial-related procedure not part of the normal medical practice.

Exclusion Criteria:

* Patients who are members of the staff of the trial center, staff of the sponsor or CRO, the investigator him/herself or close relatives of the investigator.
* Simultaneous participation in another interventional clinical trial, participation in another trial with less than 30 days or five half-lives of the IMP (whatever is longer) to screening, or previous participation in this trial.
* Ineligible for chemotherapy treatment with FOLFIRINOX or gemcitabine+Abraxane®
* Use of dronabinol or cannabis-based medicine with THC as constituent within 6 months before screening. A urine drug test will be performed during screening phase.
* Use of marihuana within the last 4 weeks and unwillingness to abstain for the duration of the study. A urine drug test will be performed during screening phase.
* Currently receiving chemotherapy or anticipated use of chemotherapy due to any condition not related to locally advanced or metastatic pancreatic cancer
* History of or existing cardiac diseases or pathological findings (e.g. chronic insufficiency NYHA III/IV, severe arrhythmia, unstable angina pectoris, myocardial infarction within the past 6 months, significant QT-prolongation etc.), which in the opinion of the investigator might interfere with the safety or tolerability of the study treatment. An ECG has to be done to exclude pathological findings and must not be older than 3 months before screening or if none is available, has to be performed during the screening phase and assessed prior to randomization
* Clinically relevant, severe pulmonary diseases, uncontrolled hypertension, or poorly controlled diabetes
* History of or existing relevant CNS and/or psychiatric disorders (e.g. schizophrenia, psychosis, manic and/or depressive disorders, suicidal ideations, etc) which might interfere with the safety or tolerability of the study treatment. Patients with reactive depression are not excluded from participation.
* Known current or past (within the last year prior to screening) alcohol, narcotics or drug abuse
* Pregnancy or breast feeding
* Known allergy to cannabinoids and other constituents of the investigational medicinal product
* Intake of prohibited concomitant medication
* Any other substantial medical condition that in the opinion of the investigator could create undue risk to the subject or could affect adherence with the trial protocol
* Legal incapacity, limited legal capacity or any other condition which makes the subject unable to understand the subject information and informed consent form (ICF)
* Patients unable or unwilling to waive driving motor vehicles or using machines especially during titration period
* Unable or unwilling to comply with the protocol regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Standardized area under the curve of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 symptom summary score over the on-treatment period. | Prior to treatment start until end of 16 weeks maintenance treatment
  The EORTC-QLQ-C30 is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The validated QLQ-C30 summary score is calculated as mean score of the 13 of the 15 EORTC QLQ-C30 scales (v3.0), based on 27 of 30 items (the Financial Impact scale and Quality of Life score are not included). A high score for a symptom scale / item (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea) represents a high level of symptomatology / problems. A high score for a functional scale (physical functioning, role functioning, cognitive functioning, emotional functioning, social functioning) represents a high / healthy level of functioning. Scores for individual items: "Not at All" = 1 point, "A Little" = 2 points, "Quite a Bit" = 3 points, "Very Much" = 4 points.
  A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.

SECONDARY OUTCOMES:
Standardized area under the curve of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 symptom summary score over the maintenance period | After 4 weeks of treatment until week 16
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The validated QLQ-C30 summary score is calculated as mean score of items. A high score for a symptom scale / item (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea) represents a high level of symptomatology / problems.
  Scores for individual items: "Not at All" = 1 point, "A Little" = 2 points, "Quite a Bit" = 3 points, "Very Much" = 4 points. A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.
Change of European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 symptom summary score from baseline to summary score over the maintenance period | From treatment start until week 16
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The validated QLQ-C30 summary score is calculated as mean score of items. A high score for a symptom scale / item (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea) represents a high level of symptomatology / problems.
  Scores for individual items: "Not at All" = 1 point, "A Little" = 2 points, "Quite a Bit" = 3 points, "Very Much" = 4 points. A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.
Symptom scales of European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 | At baseline and 2-weekly until end of treatment at week 18
  A high score for a symptom scale / item (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea) represents a high level of symptomatology / problems.
  Scores for individual items: "Not at All" = 1 point, "A Little" = 2 points, "Quite a Bit" = 3 points, "Very Much" = 4 points. A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.
Global quality of life of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 | At baseline and 2-weekly until end of treatment at week 18
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The validated QLQ-C30 summary score is calculated as mean score of items. A high score for the global health status (overall health during the past week) and global QoL (overall quality of life during the past week) represents a high QoL.
  Scores: 1 - 7, 1 = very poor and 7 = excellent. A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.
Functional scales of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 | At baseline and 2-weekly until end of treatment at week 18
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials. A high score for a functional scale (physical functioning, role functioning, cognitive functioning, emotional functioning, social functioning) represents a high / healthy level of functioning.
  Scores for individual items: "Not at All" = 1 point, "A Little" = 2 points, "Quite a Bit" = 3 points, "Very Much" = 4 points.
  A linear transformation is used to standardize the raw score, so that overall scores range from 0 to 100.
Mean change from baseline of the Glasgow Prognostic Score | At baseline and at end of treatment at week 16
  Change of serum levels of the score-defining biomarkers C-reactive protein (CRP) and albumin. Prognostic scores; 0 (CRP ≥ 10 mg/l), 1 (CRP > 10 mg/l and albumin ≥ 35 g/l), 2 CRP > 10 mg/l and albumin < 35g/l). Score 0 indicates good prognosis, score 1 intermediate prognosis and score 2 poor prognosis.
Amount of concomitant medication taken | From baseline until end of treatment at week 18
  Special focus on antiemetic, psychotropic and pain medication
Mean time to critical weight-loss (5%) | From baseline until end of treatment at week 16
  Assessed with a standard scale
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Lean body mass (LBM) | At baseline and at end of treatment at week 16
  Mean change of Lean body mass (LBM = Fat free mass FFM) kg
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Total body water (TBW) | At baseline and at end of treatment at week 16
  Mean change of Total body water (TBW) kg
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Fat mass (FM) | At baseline and at end of treatment at week 16
  Mean change of Fat mass (FM) kg
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Body cell mass (BCM) | At baseline and at end of treatment at week 16
  Mean change of Body cell mass (BCM) kg
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Extracellular mass (EM) | At baseline and at end of treatment at week 16
  Mean change of Extracellular mass (ECM) kg
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Phase angle (PA) | At baseline and at end of treatment at week 16
  Mean change of Phase angle (PA); Phase Angle has long been linked to nutritional status. This marker is fast becoming recognised as a global health marker in total body health assessment. A higher Phase Angle could mean an increase in muscle mass (body cell mass) or a decrease in fluid, either from recovery from infection or injury (a good thing!) or a decrease in fluid from dehydration (a bad thing!). A loss of fat could also increase Phase Angle.
  A lower Phase Angle could mean a loss of muscle mass (a bad thing), or an increase of fluid (rehydrating which is a good thing, or sign of inflammation or infection - a bad thing), or gaining fat (which could be a good or bad thing depending on your state of health).
  Phase Angle is a direct measurement, (not a calculation using equations) of the cell membrane.
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Resistance (Rz) | At baseline and at end of treatment at week 16
  Mean change of Resistance (Rz), unit ohm; the resistance reflects the water or fluid in the body
Mean changes from baseline for Bioelectrical Impedance Analysis (BIA) parameter Reactance(Xc) | At baseline and at end of treatment at week 16
  Mean change of Reactance (Xc), unit ohm; reactance reflects the body cell mass.
Mean change from baseline of muscle strength | At baseline and at end of treatment at week 16
  To assess physical strength of patient's handgrip strength will be measured prior and after study treatment using a hydraulic hand dynamometer; mean value of three consecutive measurements will be documented
Proportion of patients not adhering to individual baseline chemotherapy regimen | From baseline until end of treatment at week 18
  Percentage of patients who do not receive full dose of planned chemotherapy regimen and/or within scheduled time frame (interruption or delay)
Chemotherapeutic dose intensity over the treatment period of 18 weeks | From baseline until end of treatment at week 18
  The total amount of applied chemotherapy over the study treatment phase is documented
Frequency and severity of (serious) adverse events (S)AE | From baseline until safety visit at week 22
  Assessed with Common Terminology Criteria for Adverse Events (NCI-CTCAE V5.0)
Incidence of adverse drug reactions (ARs) | From baseline until safety visit at week 22
  Frequency and severity of ARs
Progression-free survival (PFS) | From treatment start until the date of first documented progression or death from any cause assessed up to week 22
  PFS in months; ; patients will be asked to agree on collection of data regarding PFS also after end of trial
Overall survival (OS) | From treatment start until death from any cause assessed up to week 22
  OS in months; ; patients will be asked to agree on collection of data regarding PFS also after end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Felix Keil, Prof.MD, Principal Investigator — Med. Dept. III, Hematolog and Oncology
Locations (11):
- Austria (8):
  - IIIrd Medical Department, Private Medical University Hospital Salzburg, Salzburg, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Abteilung für Innere Medizin IV, Wels, Upper Austria
  - Hanusch Krankenhaus der Wiener Gebietskrankenkasse, Vienna, Vienna
  - KABEG-Klinikum Klagenfurt am Woerthersee, Abteilung f. Anaesthesie u. Intensivmedizin, Klagenfurt
  - LKH Hochsteiermark - Standort Leoben Abteilung für Innere Medizin und Hämatologie und internistische Onkologie, Leoben
  - Krankenhaus d. Barmherzigen Brüder, Abt. f. Innere Medizin, Sankt Veit an der Glan
  - Pyhrn-Eisenwurzen Klinikum Steyr, Interne Medizin II, Steyr
  - KH Zams, Innere Medizin, Internistische Onkologie u. Haematologie, Zams
- Germany (3):
  - Universitätsmedizin Göttingen Abt. f. Gastroenterologie, gastrointestinale Onkologie u. Endokrinologie, Göttingen
  - München Klinik Neuperlach, München
  - Marienhospital Onkologie, Hämatologie, Palliativmedizin, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Amerongen G, Kanhai K, Baakman AC, Heuberger J, Klaassen E, Beumer TL, Strijers RLM, Killestein J, van Gerven J, Cohen A, Groeneveld GJ. Effects on Spasticity and Neuropathic Pain of an Oral Formulation of Delta9-tetrahydrocannabinol in Patients WithProgressive Multiple Sclerosis. Clin Ther. 2018 Sep;40(9):1467-1482. doi: 10.1016/j.clinthera.2017.01.016. Epub 2017 Feb 9. PMID 28189366
- [Background] Davis MP. Cannabinoids for Symptom Management and Cancer Therapy: The Evidence. J Natl Compr Canc Netw. 2016 Jul;14(7):915-22. doi: 10.6004/jnccn.2016.0094. PMID 27407130
- [Background] Cannabis-In-Cachexia-Study-Group; Strasser F, Luftner D, Possinger K, Ernst G, Ruhstaller T, Meissner W, Ko YD, Schnelle M, Reif M, Cerny T. Comparison of orally administered cannabis extract and delta-9-tetrahydrocannabinol in treating patients with cancer-related anorexia-cachexia syndrome: a multicenter, phase III, randomized, double-blind, placebo-controlled clinical trial from the Cannabis-In-Cachexia-Study-Group. J Clin Oncol. 2006 Jul 20;24(21):3394-400. doi: 10.1200/JCO.2005.05.1847. PMID 16849753
- [Background] Turgeman I, Bar-Sela G. Cannabis Use in Palliative Oncology: A Review of the Evidence for Popular Indications. Isr Med Assoc J. 2017 Feb;19(2):85-88. PMID 28457056
- [Background] Jatoi A, Windschitl HE, Loprinzi CL, Sloan JA, Dakhil SR, Mailliard JA, Pundaleeka S, Kardinal CG, Fitch TR, Krook JE, Novotny PJ, Christensen B. Dronabinol versus megestrol acetate versus combination therapy for cancer-associated anorexia: a North Central Cancer Treatment Group study. J Clin Oncol. 2002 Jan 15;20(2):567-73. doi: 10.1200/JCO.2002.20.2.567. PMID 11786587
- See also: Sponsor — http://www.agmt.at